CLINICAL TRIAL: NCT01042873
Title: The Hemodynamic Response to Prolonged Dobutamine Infusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0355-09-HMO-CTIL; 0355-09-HMO (Other: HadassahMO)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-03

CONDITIONS: Healthy; Heart Failure
Keywords: Desensitization; beta adrenergic receptors; Healthy subjects
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous dobutamine (Other): 3 hours infusion of dobutamine
  Interventions: Drug: 3 hours intravenous dobutamine

INTERVENTIONS:
Drug: 3 hours intravenous dobutamine — Intravenous dobutamine will be infused during 3 hours. At the first and last 0.5 hors of infusion dose will be increased gradually, while in the middle 2 hours dose will remain constant.

SUMMARY:
A decrease in the response of beta 1 adrenergic receptors to agonists (desensitization) is thought to play a major role in the pathogenesis of diseases such as congestive heart failure. However, currently, there is no in vivo model that will enable us to measure desensitization of the hemodynamic responses to beta 1 adrenergic receptors in vivo.

Our hypothesis is that constant 3 hours intravenous infusion of the selective beta1 adrenergic receptor agonist dobutamine will result in gradual decline in hemodynamic responses to dobutamine over time.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* consumption of any medications during the 2 weeks prior to the study
* history of chest pain or tachycardia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 3 hours

SECONDARY OUTCOMES:
Systolic blood pressure | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Bruck H, Leineweber K, Temme T, Weber M, Heusch G, Philipp T, Brodde OE. The Arg389Gly beta1-adrenoceptor polymorphism and catecholamine effects on plasma-renin activity. J Am Coll Cardiol. 2005 Dec 6;46(11):2111-5. doi: 10.1016/j.jacc.2005.08.041. Epub 2005 Nov 4. PMID 16325050